CLINICAL TRIAL: NCT04321525
Title: Psychotherapy for Young Adults With Mild-to-moderate Depression: Does Virtual Reality Increase Its Efficacy
Acronym: PSYADEP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 pandemic disrupted trial recruitment in 2020-2022. Cooperating healthcare centers lacked resources, and funding was exhausted, necessitating trial termination.
Sponsor: University of Barcelona (Other)
Collaborators: Universitat Oberta de Catalunya (Other)
Responsible Party: Principal Investigator, Dr. Guillem Feixas, full professor, University of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RTI2018-094294-B-I00
Record Dates: First submitted 2020-02-18; First posted 2020-03-25 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cognitive-behavioral therapy (CBT) (Active Comparator): Individual Cognitive Behavioral Therapy
  Interventions: Behavioral: Cognitive-behavioral therapy
- Personal construct therapy (PCT) (Experimental): Individual Personal Construct Therapy
  Interventions: Behavioral: Personal Construct Therapy
- Personal construct therapy with virtual reality (PCT-VR) (Experimental): Individual Personal Construct Therapy with an immersive virtual reality app
  Interventions: Behavioral: Personal Construct Therapy with virtual reality

INTERVENTIONS:
Behavioral: Cognitive-behavioral therapy — 10 individual one-hour sessions, with one or two booster sessions at about three months after the tenth session
  Other Names: Cognitive therapy
  Arms: Cognitive-behavioral therapy (CBT)
Behavioral: Personal Construct Therapy — 10 individual one-hour sessions, with one or two booster sessions at about three months after the tenth session
  Arms: Personal construct therapy (PCT)
Behavioral: Personal Construct Therapy with virtual reality — 10 individual one-hour sessions, with one or two booster sessions at about three months after the tenth session
  Arms: Personal construct therapy with virtual reality (PCT-VR)

SUMMARY:
Cognitive Behavioral Therapy (CBT) is the most prestigious psychological treatment for depression. However, not only do we need to increase its efficacy but also to widen the repertoire of evidence-based psychotherapeutic interventions. The importance of the patient's engagement in treatment is highlighted in the literature as a key factor for a good therapeutic outcome over and above the type of therapy. In this sense, personal construct therapy (PCT), with some promising supporting evidence, is particularly suited to fit the personal values and attitudes of each patient. In contrast to CBT, PCT does not educate patients about depression and give them directions on the changes to be made in their dysfunctional behaviors or cognitions. Rather, PCT explores their coherence with respect to the person's sense of identity, their construction of self and others, and works with the conflicts or dilemmas that appear during this conjoint exploration using the Repertory Grid Technique (RGT). In this project, for the first time, the RGT will be implemented using Virtual Reality (VR). This format could be highly appealing for young people, thus facilitating their involvement in therapy. The efficacy of this innovative application of PCT using VR (PCT-VR) will be compared to usual PCT, and to CBT in a randomized clinical trial. The Beck Depression Inventory-II is the primary outcome measure for calculating both statistical and clinical significance, but other measures will also be used at pre-, post-therapy and six-month follow up. The trial will be done in a natural health context, mostly the usual primary care center of each patient, with those who consult during the active period of the study.

Our research group has been working on both depression and personal construct theory for more than two decades (this includes our previous funded projects), particularly with a dilemma-focused intervention aimed to resolve the cognitive conflicts detected with the RGT. By fostering a technological innovation with VR, it is expected to boost the current efficacy of psychotherapy by increasing the engagement of young people and obtaining better outcomes. If these goals are met, a pathological evolution of the patient with its associated personal, health and social costs could be avoided.

DETAILED DESCRIPTION:
This project will allow to test the hypothesis that a novel brief psychotherapeutic intervention, personal construct therapy with virtual reality (PCT-VR) will be more efficacious in the treatment of mild-to-moderate depression of young adults than current treatments such as the well-established Cognitive Behavioral Therapy (CBT), and the promissory personal construct therapy (PCT). It is expected that the enhancement of a current psychotherapy with VR, based on the immersive exploration of the patient's self-identity, will increase the positive effects of existing psychological therapies (at least the other therapies included in the study) in terms of symptom reduction of depressive symptoms (primary outcome), and bettering of psychological functioning, wellbeing and satisfaction. It is assumed that the use of the VR device created for this study, will make the treatment more attractive for young adults, this increasing their engagement in the therapy process. It is hypothesized that an immersive exploration of the personal constructs used to perceive self and others will facilitate self-understanding and change. As a secondary hypothesis, it is expected that PCT, thanks to its personalized and non-prescriptive nature, will be more efficacious than CBT. Also, as reflected in the literature, it is expected that the quality of the therapeutic alliance will be associated to outcome, but whether this association varies in its intensity across therapy modalities will be also explored.

General objectives With this project, it is pursued the goal of increasing the efficacy of psychological therapies for mild-to-moderate depression in young adults. It is expected to obtain better clinical results with the promissory and novel treatment modalities (PCT and PCT-VR) than with the current most prestigious CBT. By obtaining supporting evidence for these therapies, the range of psychotherapeutic alternatives for depression will be increased and this will benefit the potential for adapting the interventions to the personal styles, characteristics and preferences of each patient. An optimal personalization of the treatment favors the patient engagement in therapy and strengthens the therapeutic alliance which, in turn, should be reflected in a facilitation of the change process.

Specific objectives

1. To assess the efficacy of an innovative VR-enhanced treatment modality of psychotherapy (PCT-VR) which has never been tested before. Differential outcomes will be considered not only in terms of statistical but also clinical significance and remission rates. In addition to the reduction of depressive symptoms our study is aimed also to better psychological functioning, wellbeing and satisfaction with the services provided.

2- To evaluate the efficacy for mild-to-moderate depression in young adults of PCT, a psychotherapeutic approach with some supporting evidence for a variety of disorders and conditions but still insufficient to be considered efficacious for depression.

3- To verify the good levels of efficacy shown by CBT in the treatment of depression, mostly in international studies.

4- To identify baseline variables predicting differential outcome such as symptom severity (also comparing mild with moderate depression), and characteristics of the personal construct system such as the level of cognitive conflict.

5- To gauge the significance of the therapeutic alliance in the different treatment modalities of the study and its influence in the therapeutic outcomes measured.

6- To explore the personal views of patients with respect to the therapy process that they will have experienced as a way to advance our knowledge of the therapy process (including potential adverse effects) of each treatment. To compare this knowledge with the quantitative results of the study might be helpful for a better understanding of the entire process.

ELIGIBILITY:
Inclusion Criteria:

* All participants will meet diagnostic criteria for mild or moderate depressive episode according to ICD-10 (current version in the Catalan health system), diagnosed using MINI, and a score above 13 and below 29 on the BDI-II questionnaire.

Exclusion Criteria:

* Patients presenting bipolar or other affective disorders (ICD-10), psychotic symptoms, substance abuse, organic brain dysfunction, acute suicidal ideation or mental retardation will be excluded from the study. The presence of other comorbid conditions (anxiety, eating or personality disorders, etc.) will not be cause for exclusion but they will be assessed and recorded and explored statistically. Finally, those who do not have enough level of competence to communicate in Spanish or Catalan, or patients with substantial visual, hearing and cognitive deficits cannot be included

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Change in Beck depression inventory second edition | BDI-II is administered at the end of therapy (10 weeks), and 6-month follow-up
  Beck Depression Inventory, Second Edition (BDI-II; Beck, Steer & Brown, 1996). It is a 21-item self-report instrument to assess the existence and severity of symptoms of depression. Both the original and the Spanish version (Sanz, Perdigón, & Vázquez, 2003) showed good psychometric properties and acceptability.

SECONDARY OUTCOMES:
Clinical Outcomes in Routine Evaluation-Outcome Measure | CORE-OM is administered at baseline, and then routinely every session (using short forms versions A and B) until the end of treatment (10 weeks), and 6-month follow-up
  Clinical Outcomes in Routine Evaluation-Outcome Measure (CORE-OM; Evans et al, 2002). It is a 34-item self-report questionnaire for the assessment of subjective wellbeing, symptoms or problems, life functioning and risk. It has good psychometric properties (Trujillo et al, 2016) and it has been adapted into Spanish for free distribution (www.ub.edu/terdep/core) . The short version (CORE-SFB) of 18 items will be used for session-to-session monitoring of the therapy process.
- Depression, Anxiety and Stress Scales | DASS-21 is administered at the end of therapy (10 weeks), and 6-month follow-up
  Depression, Anxiety and Stress Scales (DASS-21; Lovibond & Lovibond, 1995). This 21-item version of the DASS comprises 7 items for its three scales (depression, anxiety and stress) which are moderately correlated with each other. The scores for each scale range from 0 to 21. There have been studies of validation with Spanish population finding satisfactory psychometric properties (Bados, Solanas, & Andrés, 2005).
Session Rating Scale 3.0 | SRS 3.0 is administered routinely after every session, through intervention completion (10 weeks), and 6-month follow-up
  Session Rating Scale 3.0 (SRS 3.0; Duncan et al., 2003). It is a brief questionnaire designed to assess therapeutic alliance at the end of the session. It is composed of 4 items that have to be answered through a visual analog scale (VAS) of 10 centimeters. They measure the appreciation of the relationship with the therapist, agreement with the therapist about the goals and issues discussed in the session, agreement with the method or approach of the therapist, and global assessment of the session. The Spanish version obtained good levels of validity and reliability (Moggia, Niño-Robles, Miller, & Feixas, 2018)
Change Interview | administered at the end of therapy (10 weeks)
  Change Interview (Elliott, Slatick and Urman, 2001). This semi-structured interview was created to assess the changes produced throughout therapy, the useful aspects, and the adverse effects of interventions from the patient's perspective. The patient is asked about the (positive) changes he/she has experienced with the intervention, as well as the negative changes if there has been any. Questions are also asked about the attribution of such changes, and their probability of occurrence without intervention. Its functions in this study are to identify both changes that patients are aware of (in their own words) which might go unnoticed with standardized questionnaires and adverse effects (too often neglected in psychotherapy research).

OTHER OUTCOMES:
Treatment adherence scale | Administered at the end of therapy (up to 1 year)
  The Adherence to protocol scale created in a preliminary study will be used for assessing the adherence of therapists to the protocols of the assigned treatment condition. The higher the score the better the adherence in a scale from zero to ten. Two graduate students blinded to the treatment conditions and trained to use the scale reliably will rate the audiotapes of 10 sessions of CBT, PCT and PCT-VR.
Consumer Reports Effectiveness Scale | administered at the end of therapy (10 weeks)
  Consumer Reports Effectiveness Scale (CRES-4 Feixas, Pucurull, Roca, Paz, García-Grau y Bados, 2012). It consists of four items designed to evaluate whether patients are satisfied with the therapy they have received and if it has been perceived as effective or not. The total score is intended to reflect the degree of satisfaction with treatment received. To interpret CRES-4 globally, a score is considered that is on a scale ranging from 0 to 300 points. The higher the total score, the greater the effectiveness of the treatment according to the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Guillem Feixas, Ph.D, Principal Investigator — University of Barcelona
Locations (2):
- Spain (2):
  - University of Barcelona, Barcelona, Catalonia
  - Associació Centre Higiene Mental Nou Barris, Barcelona

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data for all primary and secondary outcomes, after deidentification
Supporting Information: Study Protocol
Time Frame: Data will be available after six months of study completion
Access Criteria: Researchers who provide a methodologically sound proposal whose proposed use of the data has been approved by an independent review committee

REFERENCES:
- [Background] Montesano A, Medina JC, Paz C, Garcia-Mieres H, Nino-Robles N, Garcia-Grau E, Crespillo JC, Garcia-Gutierrez A, Alabernia-Segura M, Feixas G. Does virtual reality increase the efficacy of psychotherapy for young adults with mild-to-moderate depression? A study protocol for a multicenter randomized clinical trial. Trials. 2021 Dec 13;22(1):916. doi: 10.1186/s13063-021-05809-1. PMID 34903251